CLINICAL TRIAL: NCT00701415
Title: A Randomized, Multicenter, Multinational, Phase 3B, Open-Label, Parallel-Group Study of Fabrazyme (Agalsidase Beta) in Treatment-Naïve Male Pediatric Patients With Fabry Disease Without Severe Symptoms
Brief Title: A Study of Two Fabrazyme (Agalsidase Beta) Dosing Regimens in Treatment-naïve, Male Pediatric Patients Without Severe Symptoms
Acronym: FIELD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGAL06207; 2007-005668-28 (EudraCT Number); EFC12821 (Other: Sanofi)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Fabry Disease
Keywords: α-GAL, α-Galactosidase-A, r-hαGAL
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fabrazyme 0.5 mg/kg (Experimental): Fabrazyme 0.5 mg/kg was administered every 2 weeks (up to 131 infusion) up to 260 weeks, the total infusion time was not less than 45 minutes. In case of significant progression of Fabry disease, the dose was increased to 1.0 mg/kg every 2 weeks.
  Interventions: Biological: Agalsidase beta
- Fabrazyme 1.0 mg/kg (Experimental): Fabrazyme 1.0 mg/kg was administered every 4 weeks (up to 66 infusion) up to 260 weeks, the total infusion time was not less than 90 minutes. In case of significant progression of Fabry disease, the dose was increased to 1.0 mg/kg every 2 weeks.
  Interventions: Biological: Agalsidase beta

INTERVENTIONS:
Biological: Agalsidase beta — Powder for concentrate for solution for infusion 1.0 mg/kg/4 weeks
  Other Names: Fabrazyme; Recombinant human α-galactosidase A (r-hαGAL)
  Arms: Fabrazyme 0.5 mg/kg
Biological: Agalsidase beta — Powder for concentrate for solution for infusion 0.5 mg/kg/2 weeks
  Other Names: Fabrazyme; Recombinant human α-galactosidase A (r-hαGAL)
  Arms: Fabrazyme 1.0 mg/kg

SUMMARY:
The purpose of this study was to determine whether 2 alternative dosing regimens of Fabrazyme (Agalsidase beta) (1.0 mg/kg every 4 weeks or 0.5 mg/kg every 2 weeks) were effective in treatment-naïve pediatric participants without severe symptoms. Participants were to be treated for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The participant and/or participant's parent(s)/legal guardian(s) must provide written informed assent/consent prior to any protocol-related procedures being performed.
* The participant must had a confirmed diagnosis of Fabry disease as documented by leukocyte α-Galactosidase A (αGAL) activity of <4 nmol/hr/mg leukocyte (preferred assay; resulted from a central laboratory). If the leukocyte αGAL activity assay was difficult to obtain, the participant might be enrolled based on documented plasma αGAL <1.5 nmol/hr/mL, with the agreement of the Medical Monitor (resulted from a central laboratory).
* The participant must had evidence of globotriaosylceramide (GL-3) accumulation as documented by plasma GL-3 (>7.0 µg/mL) or urinary GL-3 (>0.3 mg GL-3/mmol creatinine) levels (results from a central laboratory).
* The participant must be male ≥5 and ≤18 years of age.

Exclusion Criteria:

* Participant had albuminuria (first morning void urinary albumin/creatinine ratio >30 mg/g on at least 2 out of 3 consecutive samples, each at least 1 week apart).
* Participant had a Glomerular Filtration Rate (GFR) by iohexol <90 L/min/1.73m^2. In case of properly documented low protein intake, values as low as 80 mL/min/1.73 m^2 might be acceptable, after consultation with the Medical Monitor.
* Participant had documented evidence of stroke or transient ischemic attack (TIA), or if a brain magnetic resonance imaging (MRI) had been performed, bright lesions >2 mm on T2- or fluid attenuated inversion recovery (FLAIR)- weighted images within the white matter or the basal ganglia.
* Participant had severe and recurrent acroparesthesia, judged by the physician as frequent (more than once a week) pain episodes for at least 3 months that influenced daily activities, irrespective of medication.
* Participant had an end-diastolic left ventricular posterior wall thickness (LVPWTd) and/or an end-diastolic interventricular septum thickness (IVSTd)≥2 standard deviations (SD) compared to normal (based on body surface area [BSA] normal ranges from Kampmann, et al 2000) as read at the study site.
* Participant had received prior treatment specific to Fabry Disease.
* Participant had participated in a study employing an investigational drug within 30 days of the start of their participation in this study.
* Participant had any medical condition or extenuating circumstance, which in the opinion of the Study Investigator, could interfere with study compliance.
* Participant had any medical condition or extenuating circumstance, for example diabetes mellitus, which in the opinion of the Study Investigator, could interfere with the interpretation of study results.
* Participant was on treatment with angiotensin converting enzyme inhibitors/angiotensin receptor blockers (ACEIs/ARBs).
* Participant had any contra-indication mentioned in the labeling of Fabrazyme and/or iohexol (Omnipaque).
* Participant or parent(s)/legal guardian(s) was unwilling to comply with the requirements of the protocol.

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (12):
- United States (3):
  - Decatur, Georgia
  - Cincinnati, Ohio
  - Seattle, Washington
- Buenos Aires, Argentina
- Passo Fundo, Rio Grande do Sul, Brazil
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, QC
- Prague, Czechia
- Amsterdam, Netherlands
- Bergen, Norway
- Warsaw, Poland
- Cambridge, United Kingdom

REFERENCES:
- [Derived] Wijburg FA, Benichou B, Bichet DG, Clarke LA, Dostalova G, Fainboim A, Fellgiebel A, Forcelini C, An Haack K, Hopkin RJ, Mauer M, Najafian B, Scott CR, Shankar SP, Thurberg BL, Tondel C, Tylki-Szymanska A, Ramaswami U. Characterization of early disease status in treatment-naive male paediatric patients with Fabry disease enrolled in a randomized clinical trial. PLoS One. 2015 May 8;10(5):e0124987. doi: 10.1371/journal.pone.0124987. eCollection 2015. PMID 25955246
- [Derived] Rombach SM, Smid BE, Bouwman MG, Linthorst GE, Dijkgraaf MG, Hollak CE. Long term enzyme replacement therapy for Fabry disease: effectiveness on kidney, heart and brain. Orphanet J Rare Dis. 2013 Mar 25;8:47. doi: 10.1186/1750-1172-8-47. PMID 23531228

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 sites in 9 countries. A total of 44 participants were screened between 17 June 2008 and 12 April 2010.
Pre-assignment Details: Of 44 screened participants, 31 were randomized in 1:1 ratio to fabrazyme 0.5 mg/kg and fabrazyme 1.0 mg/kg within each age stratum (5 to ≤11 years [children] and 12 to ≤18 years [adolescents]). 13 participants were screen failure due to failure to meet inclusion criteria or withdrawal of consent prior to all screening assessments being completed.
Groups:
- Fabrazyme 0.5 mg/kg: Fabrazyme 0.5 mg/kg was administered every 2 weeks (up to 131 infusions) up to 260 weeks, the total infusion time was not less than 45 minutes. In case of significant progression of Fabry disease, the dose was increased to 1.0 mg/kg every 2 weeks.
- Fabrazyme 1.0 mg/kg: Fabrazyme 1.0 mg/kg was administered every 4 weeks (up to 66 infusions) up to 260 weeks, the total infusion time was not less than 90 minutes. In case of significant progression of Fabry disease, the dose was increased to 1.0 mg/kg every 2 weeks.
Period: Overall Study
Arm/Group | Fabrazyme 0.5 mg/kg | Fabrazyme 1.0 mg/kg
Started | 16 | 15
Completed | 15 | 14
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Social/family issues and needle phobia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fabrazyme 0.5 mg/kg | Fabrazyme 1.0 mg/kg | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (4) | 11.9 (4.5) | 11.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Skin Globotriaosylceramide (GL-3) Clearance From Superficial Skin Capillary Endothelium
Description: Skin biopsies were taken at Baseline, Week 52, Week 156 and Week 260 or early withdrawal and analyzed for cellular GL-3 accumulation (inclusions) by light microscopy. Each biopsy was scored for GL-3 accumulation on a severity score-scale of none, mild, moderate, severe (0-1-2-3). Scores are categorized as normal (score = 0) or abnormal (score = 1, 2 or 3). Data was summarized in terms of number of participants with none/trace, mild, moderate and severe biopsy scores.
Time Frame: Baseline, Week 52, Week 156 and Week 260
Population: Analysis was performed on Full analysis set (FAS), which included all randomized participants who received at least 1 infusion of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Fabrazyme 0.5 mg/kg | Fabrazyme 1.0 mg/kg
Number analyzed (Participants) | 16 | 15
Percentage of participants
  Zero (0) Skin GL-3 Score at Baseline | 18.8 | 33.3
  Zero (0) Skin GL-3 Score at Week 52 | 75 | 80
  Zero (0) Skin GL-3 Score at Week 156 | 56.3 | 80
  Zero (0) Skin GL-3 Score at Week 260 | 68.8 | 66.7
  Mild (1) Skin GL-3 Score at Baseline | 6.3 | 0
  Mild (1) Skin GL-3 Score at Week 52 | 6.3 | 13.3
  Mild (1) Skin GL-3 Score at Week 156 | 18.8 | 0
  Mild (1) Skin GL-3 Score at Week 260 | 12.5 | 20
  Moderate (2) Skin GL-3 Score at Baseline | 75 | 66.7
  Moderate (2) Skin GL-3 Score at Week 52 | 0 | 0
  Moderate (2) Skin GL-3 Score at Week 156 | 6.3 | 13.3
  Moderate (2) Skin GL-3 Score at Week 260 | 0 | 6.7
  Severe (3) Skin GL-3 Score at Baseline | 0 | 0
  Severe (3) Skin GL-3 Score at Week 52 | 0 | 0
  Severe (3) Skin GL-3 Score at Week 156 | 0 | 0
  Severe (3) Skin GL-3 Score at Week 260 | 0 | 0
  Missing Skin GL-3 Score at Baseline | 0 | 0
  Missing Skin GL-3 Score at Week 52 | 18.8 | 6.7
  Missing Skin GL-3 Score at Week 156 | 18.8 | 6.7
  Missing Skin GL-3 Score at Week 260 | 18.8 | 6.7

2. Secondary Outcome: Percent Change From Baseline in GL-3 Clearance From Plasma
Description: Plasma samples were assayed for GL-3 clearance using a validated tandem mass spectrometry with an upper limit of normal plasma GL-3 level of 7.0 μg/mL. Number of participants analyzed=participants with both baseline and post-baseline GL-3 plasma clearance assessment. Here 'n' signifies number of participants with available data for specified category.
Time Frame: Baseline, Week 12, 28, 40, 52, 80, 104, 132, 156, 184, 208, 236 and 260
Population: Analysis was performed on FAS.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Fabrazyme 0.5 mg/kg | Fabrazyme 1.0 mg/kg
Number analyzed (Participants) | 14 | 14
Percent change
  Week 12 (n=14, 11) | -52.37 (10.12) | -52.74 (6.79)
  Week 28 (n=14, 14) | -49.06 (15.43) | -47.55 (16.75)
  Week 40 (n=13, 14) | -52.01 (11.29) | -50.82 (12.87)
  Week 52 (n=14, 14) | -52.29 (10.48) | -45.87 (16.01)
  Week 80 (n=13, 14) | -52.91 (13.93) | -48.93 (14.75)
  Week 104 (n=13, 14) | -51.08 (20.45) | -39.92 (18.69)
  Week 132 (n=11, 14) | -61.39 (10.71) | -52.97 (17.1)
  Week 156 (n=11, 14) | -48.72 (18.48) | -44.83 (14.14)
  Week 184 (n=12, 14) | -53.62 (19.38) | -49.08 (17.93)
  Week 208 (n=12, 14) | -48.83 (16.80) | -46.09 (16.84)
  Week 236 (n=12, 14) | -56.44 (12.08) | -47.25 (13.04)
  Week 260 (n=11, 14) | -59.95 (12.39) | -46.34 (14.01)

3. Secondary Outcome: Percent Change From Baseline in GL-3 Clearance From Urine
Description: Plasma samples were assayed for total urine GL-3 clearance using a validated tandem mass spectrometry with an upper limit of normal of <0.030 mg/mmoL of creatinine. Number of participants analyzed=participants with both baseline and post-baseline GL-3 urine clearance assessment. Here 'n' signifies number of participants with available data for specified category.
Time Frame: Baseline, Week 12, 28, 40, 52, 80, 104, 132, 156, 184, 208, 236 and 260
Population: Analysis was performed on FAS.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Fabrazyme 0.5 mg/kg | Fabrazyme 1.0 mg/kg
Number analyzed (Participants) | 15 | 15
Percent change
  Week 12 (n=15, 14) | -50.77 (64.59) | -63.39 (38.81)
  Week 28 (n=15, 15) | -50.84 (100.61) | -52.55 (58.59)
  Week 40 (n=15, 14) | -44.22 (105.03) | -63.87 (24.41)
  Week 52 (n=15, 14) | -70.1 (41.4) | -20.72 (156.1)
  Week 80 (n=14, 14) | -35.84 (102.31) | 35.22 (238.61)
  Week 104 (n=14, 14) | -21.92 (138.78) | -56.39 (42.39)
  Week 132 (n=13, 14) | -48.79 (100.1) | -45.61 (48.84)
  Week 156 (n=13, 14) | -65.57 (52.11) | -28.92 (84.32)
  Week 184 (n=13, 14) | -76.54 (38.93) | -10.5 (146.86)
  Week 208 (n=13, 14) | -60.94 (67.99) | -50.93 (46.52)
  Week 236 (n=13, 14) | -69.08 (51.72) | -40.09 (77.04)
  Week 260 (n=13, 14) | -57.59 (93.74) | -28.27 (56.79)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 264) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (the time from the first infusion of the study drug up to 28 days after the last infusion of study drug). Safety population included all randomized participants who received at least one infusion of Fabrazyme.
Arm/Group | Fabrazyme 0.5 mg/kg | Fabrazyme 1.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 6/16 | 5/15
Other Adverse Events (participants affected / at risk) | 16/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme 0.5 mg/kg (N=16) | Fabrazyme 1.0 mg/kg (N=15)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 1
CELLULITIS (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1
OTITIS MEDIA (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1
TINEA PEDIS (Infections and infestations) | 0 | 1
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
BODY MASS INDEX DECREASED (Investigations) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 1
TREMOR (Nervous system disorders) | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0
MICROALBUMINURIA (Renal and urinary disorders) | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
CENTRAL VENOUS CATHETERISATION (Surgical and medical procedures) | 1 | 0
ELECTIVE SURGERY (Surgical and medical procedures) | 1 | 0
CHILLS (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme 0.5 mg/kg (N=16) | Fabrazyme 1.0 mg/kg (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 2
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 | 0
MONOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 2 | 1
CONDUCTIVE DEAFNESS (Ear and labyrinth disorders) | 1 | 2
DEAFNESS (Ear and labyrinth disorders) | 1 | 0
DEAFNESS BILATERAL (Ear and labyrinth disorders) | 1 | 0
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 | 0
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 | 2
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 0 | 1
OTORRHOEA (Ear and labyrinth disorders) | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 3 | 4
TYMPANIC MEMBRANE HYPERAEMIA (Ear and labyrinth disorders) | 1 | 0
HYPERPARATHYROIDISM SECONDARY (Endocrine disorders) | 1 | 1
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 2
CORNEAL DEPOSITS (Eye disorders) | 1 | 0
DRY EYE (Eye disorders) | 1 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 1
OCULAR VASCULAR DISORDER (Eye disorders) | 0 | 1
PHOTOPHOBIA (Eye disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 0 | 1
VISUAL ACUITY REDUCED (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 | 6
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 4
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
DENTAL CARIES (Gastrointestinal disorders) | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 10 | 8
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 1
FOOD POISONING (Gastrointestinal disorders) | 1 | 0
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 2 | 1
NAUSEA (Gastrointestinal disorders) | 9 | 7
ORAL MUCOSAL ERYTHEMA (Gastrointestinal disorders) | 0 | 1
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 9 | 7
ASTHENIA (General disorders) | 3 | 1
CATHETER SITE PAIN (General disorders) | 0 | 1
CHEST DISCOMFORT (General disorders) | 0 | 2
CHILLS (General disorders) | 6 | 2
FACE OEDEMA (General disorders) | 2 | 0
FATIGUE (General disorders) | 5 | 2
FEELING COLD (General disorders) | 3 | 1
FEELING HOT (General disorders) | 0 | 3
FEELING OF BODY TEMPERATURE CHANGE (General disorders) | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 0
INFUSION SITE PAIN (General disorders) | 1 | 0
INJECTION SITE HAEMORRHAGE (General disorders) | 1 | 0
MALAISE (General disorders) | 2 | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 3 | 2
PAIN (General disorders) | 4 | 3
PYREXIA (General disorders) | 12 | 8
SOFT TISSUE INFLAMMATION (General disorders) | 0 | 1
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 1
CATHETER SITE INFECTION (Infections and infestations) | 0 | 1
CHLAMYDIAL INFECTION (Infections and infestations) | 0 | 1
CONJUNCTIVITIS (Infections and infestations) | 0 | 1
COXSACKIE VIRAL INFECTION (Infections and infestations) | 1 | 0
EAR INFECTION (Infections and infestations) | 5 | 1
ENTEROBIASIS (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 2 | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 3 | 1
HERPES SIMPLEX (Infections and infestations) | 1 | 1
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 1
IMPETIGO (Infections and infestations) | 2 | 1
INFLUENZA (Infections and infestations) | 3 | 3
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
MOLLUSCUM CONTAGIOSUM (Infections and infestations) | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 7 | 5
ORAL HERPES (Infections and infestations) | 2 | 0
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 | 1
PARASITIC GASTROENTERITIS (Infections and infestations) | 0 | 1
PHARYNGITIS (Infections and infestations) | 2 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 0
RHINITIS (Infections and infestations) | 5 | 3
SINUSITIS (Infections and infestations) | 3 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
TINEA INFECTION (Infections and infestations) | 0 | 1
TINEA VERSICOLOUR (Infections and infestations) | 1 | 0
TONSILLITIS (Infections and infestations) | 1 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 5
VIRAL INFECTION (Infections and infestations) | 2 | 1
VIRAL PHARYNGITIS (Infections and infestations) | 0 | 1
VIRAL RHINITIS (Infections and infestations) | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 2
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 2 | 1
EAR INJURY (Injury, poisoning and procedural complications) | 0 | 1
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
FROSTBITE (Injury, poisoning and procedural complications) | 1 | 0
GENITAL INJURY (Injury, poisoning and procedural complications) | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 1
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 2
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 1
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 | 1
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 | 1
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
BETA 2 MICROGLOBULIN INCREASED (Investigations) | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 0 | 1
BODY TEMPERATURE INCREASED (Investigations) | 0 | 1
EOSINOPHIL COUNT INCREASED (Investigations) | 1 | 0
HEART RATE INCREASED (Investigations) | 0 | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 1 | 1
URINE ALBUMIN/CREATININE RATIO ABNORMAL (Investigations) | 1 | 0
VITAMIN B12 DECREASED (Investigations) | 0 | 2
VITAMIN D DECREASED (Investigations) | 1 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
OBESITY (Metabolism and nutrition disorders) | 0 | 1
UNDERWEIGHT (Metabolism and nutrition disorders) | 1 | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 5
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BURNING SENSATION (Nervous system disorders) | 1 | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 4 | 4
DYSGEUSIA (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 8 | 4
MIGRAINE (Nervous system disorders) | 1 | 1
PARAESTHESIA (Nervous system disorders) | 6 | 3
PRESYNCOPE (Nervous system disorders) | 2 | 1
SLOW RESPONSE TO STIMULI (Nervous system disorders) | 1 | 0
SPEECH DISORDER (Nervous system disorders) | 0 | 1
TREMOR (Nervous system disorders) | 1 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 1 | 0
DISORIENTATION (Psychiatric disorders) | 1 | 0
DYSPHORIA (Psychiatric disorders) | 1 | 0
HALLUCINATION (Psychiatric disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 2 | 0
LISTLESS (Psychiatric disorders) | 1 | 0
PANIC ATTACK (Psychiatric disorders) | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 2 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
HYDROURETER (Renal and urinary disorders) | 1 | 0
MICROALBUMINURIA (Renal and urinary disorders) | 0 | 1
PENILE DISCHARGE (Reproductive system and breast disorders) | 0 | 1
PENILE PAIN (Reproductive system and breast disorders) | 0 | 1
SCROTAL ANGIOKERATOMA (Reproductive system and breast disorders) | 2 | 1
ALLERGIC COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ALLERGIC RESPIRATORY SYMPTOM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 5
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 5 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 6
PHARYNGEAL ERYTHEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACNE (Skin and subcutaneous tissue disorders) | 1 | 0
ANGIOKERATOMA (Skin and subcutaneous tissue disorders) | 9 | 5
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1
MILIARIA (Skin and subcutaneous tissue disorders) | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 1
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 4 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | 2 | 1
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 0 | 1
UMBILICAL ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1
SINUS OPERATION (Surgical and medical procedures) | 1 | 0
ANGIOPATHY (Vascular disorders) | 0 | 1
FLUSHING (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 1
PALLOR (Vascular disorders) | 2 | 1
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0
INFUSION SITE EXTRAVASATION (General disorders) | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
PROTEIN URINE PRESENT (Investigations) | 1 | 0
CATARRH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0
PERIORBITAL OEDEMA (Eye disorders) | 1 | 0
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 | 0
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 2
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
HORDEOLUM (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.